CLINICAL TRIAL: NCT02621619
Title: Randomized Clinical Trial of IV Acetaminophen as an Analgesic Adjunct to IV Hydromorphone in the Treatment of Acute Severe Pain in Elderly ED Patients
Brief Title: IV Acetaminophen as an Analgesic Adjunct
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Andrew Chang, MD, Professor of Emergency Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-5369; 7K23AG033100-07 (NIH)
Record Dates: First submitted 2015-11-21; First posted 2015-12-03 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Acute Pain
Keywords: Older adults; Elderly; Acute pain; IV acetaminophen; IV hydromorphone; Analgesia; Adjunctive analgesia
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Acetaminophen; Hydromorphone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- IV acetaminophen + 0.5 mg IV hydromorphone (Experimental): 1 gram IV acetaminophen in addition to 0.5 mg IV hydromorphone
  Interventions: Drug: IV acetaminophen + 0.5 mg IV hydromorphone
- Normal saline + 0.5 mg IV hydromorphone (Placebo Comparator): 100 ml normal saline placebo in addition to 0.5 mg IV hydromorphone
  Interventions: Drug: Normal saline + 0.5 mg IV hydromorphone

INTERVENTIONS:
Drug: IV acetaminophen + 0.5 mg IV hydromorphone — 1 gram (100 ml) IV acetaminophen in addition to 0.5 mg IV hydromorphone
  Other Names: Ofirmev
  Arms: IV acetaminophen + 0.5 mg IV hydromorphone
Drug: Normal saline + 0.5 mg IV hydromorphone — 100 cc normal saline placebo in addition to 0.5 mg IV hydromorphone
  Other Names: Placebo
  Arms: Normal saline + 0.5 mg IV hydromorphone

SUMMARY:
To determine the efficacy of intravenous (IV) acetaminophen as an analgesic adjunct to IV hydromorphone in the treatment of acute severe pain in the elderly Emergency Department (ED) patients.

DETAILED DESCRIPTION:
A randomized controlled trial to determine the efficacy of 1 gram IV acetaminophen as an analgesic adjunct to 0.5 mg IV hydromorphone in the treatment of acute severe pain in the elderly ED patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute (less than 1 week in duration) severe pain necessitating use of intravenous (IV) opioids in the judgement of the treating attending physician

Exclusion Criteria:

* Use of other opioids or tramadol within past 24 hours: to avoid introducing assembly bias related to recent opioid use, since this may affect baseline levels of pain and need for analgesics.
* Prior adverse reaction to hydromorphone, morphine, or acetaminophen.
* Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in modulation of pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
* Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter pain perception.
* Systolic Blood Pressure (SBP) <100 mm Hg: Opioids can produce peripheral vasodilation that may result in orthostatic hypotension.
* Heart Rate (HR) < 60/min: Opioids can cause bradycardia.
* Oxygen saturation < 95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
* Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
* Patients using transdermal pain patches

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, MD, MS, Principal Investigator — Albany Medical College
Locations (1):
- Montefiore Medical Center Moses Division Emergency Department, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Acetaminophen + 0.5 mg IV Hydromorphone: 1 gram IV acetaminophen in addition to 0.5 mg IV hydromorphone
  IV acetaminophen + 0.5 mg IV hydromorphone: 1 gram (100 ml) IV acetaminophen in addition to 0.5 mg IV hydromorphone
  0.5 mg IV hydromorphone: Both groups (intervention and placebo) will receive 0.5 mg IV hydromorphone
- Placebo + 0.5 mg IV Hydromorphone: 100 ml normal saline placebo in addition to 0.5 mg IV hydromorphone
  Normal saline + 0.5 mg IV hydromorphone: 100 cc normal saline placebo in addition to 0.5 mg IV hydromorphone
  0.5 mg IV hydromorphone: Both groups (intervention and placebo) will receive 0.5 mg IV hydromorphone
Period: Overall Study
Arm/Group | IV Acetaminophen + 0.5 mg IV Hydromorphone | Placebo + 0.5 mg IV Hydromorphone
Started | 80 | 79
Completed | 80 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen + 0.5 mg IV Hydromorphone | Placebo + 0.5 mg IV Hydromorphone | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [69 to 79] | 72 [68 to 77] | 72 [69 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 50 | 48 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 51 | 51 | 102
  African American | 20 | 12 | 32
  White | 7 | 13 | 20
  Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 80 | 79 | 159
Baseline Pain intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS) from 0 (no pain) to 10 (worst pain imaginable).
  This baseline measure indicates the number of participants reporting a given NRS score.
  Participants
    5-7 | 13 | 10 | 23
    8 | 14 | 24 | 38
    9 | 14 | 8 | 22
    10 | 17 | 18 | 35
Number of patients nauseated before receiving study medication [Count of Participants; unit: Participants] — Number of patients nauseated due to their condition, whether as a symptom on its own or due to their level of pain. Those experiencing nausea or vomiting at baseline would not be counted with those who experience nausea or vomiting as a side effect of study medication when comparing the effects and side effects of the study medication.
  Participants
    Yes - Nauseated | 34 | 38 | 72
    No - not nauseated | 46 | 41 | 87
Number of patients vomited before receiving study medication [Count of Participants; unit: Participants] — Number of patients vomiting due to their condition, whether as a symptom on its own or due to their level of pain. Those experiencing nausea or vomiting at baseline would not be counted with those who experience nausea or vomiting as a side effect of study medication when comparing the effects and side effects of the study medication.
  Participants
    Yes - Vomited | 17 | 18 | 35
    No - Did not vomit | 63 | 61 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity, Baseline to 60 Minutes After Medication Infused
Description: Pain intensity is measured on the numerical rating scale (NRS) from 0 (no pain) to 10 (worst pain imaginable).
  Change in pain intensity is calculated by subtracting pain intensity at 60 minutes from pain intensity at baseline [e.g. Change = NRS(baseline) - NRS(60 min)].
  Note that a positive change number indicates that pain score decreased after medication was given, while a negative change number indicates that pain score increased after medication was given.
Time Frame: baseline and 60 minutes after medication was infused
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Acetaminophen + 0.5 mg IV Hydromorphone | Placebo + 0.5 mg IV Hydromorphone
Number analyzed (Participants) | 80 | 79
units on a scale | 5.8 (3.2) | 5.2 (3.0)

2. Secondary Outcome: Change in Pain Intensity Over Time
Description: Pain intensity is measured on the numerical rating scale from 0 (no pain) to 10 (worst pain imaginable).
  Change in pain intensity is calculated by subtracting pain intensity at a later time point from pain intensity at baseline [e.g. Change = NRS(baseline) - NRS(15 min)].
  Change over time is from baseline to a series of time points: 5 minutes, 15 minutes, 30 minutes, and 45 minutes
Time Frame: baseline to 5 min, 15 min, 30 min, and 45 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Acetaminophen + 0.5 mg IV Hydromorphone | Placebo + 0.5 mg IV Hydromorphone
Number analyzed (Participants) | 80 | 79
units on a scale
  Baseline to 5 minutes | 3.4 (2.8) | 2.9 (2.4)
  Baseline to 15 minutes | 4.7 (3.1) | 4.0 (2.6)
  Baseline to 30 minutes | 5.1 (2.9) | 4.8 (2.6)
  Baseline to 45 minutes | 5.5 (2.9) | 5.2 (2.8)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | IV Acetaminophen + 0.5 mg IV Hydromorphone | Placebo + 0.5 mg IV Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/79
Other Adverse Events (participants affected / at risk) | 16/80 | 13/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IV Acetaminophen + 0.5 mg IV Hydromorphone (N=80) | Placebo + 0.5 mg IV Hydromorphone (N=79)
Nausea (Gastrointestinal disorders) | 8/46 | 8/41 — Only includes patients who were neither nauseated or vomiting before receiving study medication. Those with symptoms before medication infusion were not experiencing the symptom as a side effect, and were therefore not included
Vomiting (Gastrointestinal disorders) | 2/46 | 1/41 — Only includes patients who were neither nauseated or vomiting before receiving study medication. Those with symptoms before medication infusion were not experiencing the symptom as a side effect, and were therefore not included
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Heart rate < 50 beats/min (Cardiac disorders) | 1 | 0
Oxygen saturation < 95% (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Systolic blood pressure < 90 mmHg (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02621619/Prot_SAP_000.pdf